CLINICAL TRIAL: NCT02889172
Title: Brief Intervention for Reducing Depressive and Anxiety Symptoms and Their Impact on Metabolic Variables in Patients With Type II Diabetes Mellitus and Obesity
Brief Title: Intervention for Reducing Psychiatric Symptoms and Metabolic Variables in Patients With Diabetes Mellitus (DM)
Acronym: DM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Valerio Villamil-Salcedo, PhD, Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SC-14-2411
Record Dates: First submitted 2015-04-30; First posted 2016-09-05 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Problem Solving Therapy (Experimental): Will be apply a Brief Intervention (PST) for patients with Type II Diabetes Mellitus and Obesity who receive treatment in primary care centers from Mexico City. The aim is evaluate if PST improvement the depressive and anxiety symptoms and help to adhere to treatment and stabilize their metabolic variables
  Interventions: Behavioral: Problem Solving Therapy
- Control (No Intervention): This group will receive the usual treatment , without intervention with Brief Intervention ( PST )

INTERVENTIONS:
Behavioral: Problem Solving Therapy — It will be apply a Brief Intervention (PST) for patients with Type II Diabetes Mellitus and Obesity who receive treatment in primary care centers from Mexico City to evaluate if PST improvement the depressive and anxiety symptoms and help to adhere to treatment and stabilize their metabolic variables
  Arms: Problem Solving Therapy

SUMMARY:
The purpose of this study is apply a Brief Intervention (PST) in Diabetic and Obesity patient in primary care of Mexico City to improve their depressive and anxious symptoms and stabilization of metabolic variables.

DETAILED DESCRIPTION:
Diabetes and depression are chronic diseases that affect the quality of life of people and they increase disability and reduced life expectancy. The World Health Organization estimates there will be 300 million people with diabetes worldwide. The International Diabetes Federation warns that there are currently 382 million diabetics and may increase to 471 million in 2035 if it fails to make an international preventive action.

Furthermore, depression and anxiety disorders are the most common mental disorders worldwide. It is estimated that in 2030, depression will be the principal cause of all diseases worldwide; while anxiety disorders are related to other mental and medical conditions that prolong disability.

For these reasons, researchers have developed brief psychotherapeutic treatments with good results (Cognitive and Behavioural Therapy, Interpersonal therapy, and others) but with limitations due to lack of trained personnel for such interventions. However, the need for the care of people with diabetes with depression and anxiety symptoms are increasing, and pharmacological and therapeutic treatments are not enough. In other countries are using the Problem Solving Therapy (PST) as a brief technique to support the patient for possible solutions for daily problems which will generate emotional distress and depressive and anxiety symptoms. PST focuses on learning to cope with specific problems areas and where therapist and patient work collaboratively to identify and prioritise key problem areas, to break problems down into specific, manageable tasks, problem solve, and develop appropriate coping behaviours for problems. World Health Organization recommends the PST for depression treatment, which act "in the here and now" that helps identify a relationship between physical and emotional symptoms. Previous studies have shown the efficacy of the PST in reducing depressive and anxiety symptoms. The therapist may be a general practitioner, nurse, psychologist, social worker, etc., which serves as "advisor or counselor" while the patient is an active entity to solve their problems.

Objective The aim of this study is apply a Brief Intervention (PST) in Diabetic and Obesity patients in primary care centers of Mexico City to improve their depressive and anxious symptoms and assess their impact on treatment and stabilization of metabolic variables.

Method First Stage: Training medical students who are in last part of their education of medicine.

Second Stage: Application of brief intervention (PST) in patients with diagnosis of Diabetes and Obesity.

Stage Three: Analysis of results and publication of the study. Study design. A randomized, longitudinal, comparative clinical trial will be used.

Patients:

The study population will be 70 patients (35 experimental and 35 controls) of 11 primary care centers in Mexico City, with diagnosis of type II diabetes mellitus and / or obesity.

Inclusion criteria

1. 35-70 years old
2. Female and male
3. Type II Diabetes Mellitus
4. Obesity (BMI ≥ 30)
5. K-10 ≥ 21 points
6. Beck Depression Inventory 13 to ≤ 28 points
7. Beck Anxiety Inventory 7 to ≤ 25 points
8. Informed consent accepted and signed

Exclusion criteria

1. Severe depression or suicidal ideation
2. Type I Diabetes Mellitus

Procedure. Patients with K-10 ≥ 21 will invited to participate in the project; sign the informed consent and complete the Depression and Anxiety Beck Inventory; randomly, each subject will be assigned to the experimental or control group. Patients in the experimental group will receive the PST while the control group will receive usual treatment.

Metabolic variables: Glucose, weight, blood pressure, body mass index, total cholesterol, triglycerides and waist circumference at baseline, at 6 weeks and 4 months will be evaluated during the study.

Statistical Analysis. Percentages, means, standard deviation, Chi square, t student for independent samples and analysis of variance for repeated measures will be used.

ELIGIBILITY:
Inclusion Criteria:

1. 35-70 years old
2. Female and male
3. Type II Diabetes Mellitus
4. Obesity (BMI ≥ 30)
5. K-10 ≥ 21 points
6. Beck Depression Inventory 13 to ≤ 28 points
7. Beck Anxiety Inventory 7 to ≤ 25 points
8. Informed consent accepted and signed

Exclusion Criteria:

1. Severe depression or suicidal ideation
2. Type I Diabetes Mellitus

Elimination criteria

1. Questionnaires and scales incomplete
2. Two sessions of PST missing
3. Exacerbation of depressive and / or anxious symptoms during the intervention or monitoring

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-02; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | Six months
  The Beck Depression Inventory is a questionnaire of 21 items , is a self- applied instrument ; and determines the severity of depression in a Likert scale ranging from 0 to 4 points ; the minimum score is 0 and the maximum of 63 points : 0-13 = minimal depression ; 14-19 = mild depression ; 20-28 = moderate depression ; 29-63 = severe depression .
  This instrument has been used in several international studies and in Mexico showing validity and reliability.

SECONDARY OUTCOMES:
Beck Anxiety Inventory | Six Months
  The Beck Anxiety Inventory is a semi-structured questionnaire, which applies as assessed clinical having the patient. It consists of 21 questions Likert from 0 to 4 points that assesses the severity of anxiety : 0-7 = minimal anxiety ; 8-15 = mild anxiety ; 16-25 = moderate anxiety ; 26-63 = severe anxiety. The questionnaire has been validated in international studies in Mexico and in clinical settings .
Simplified Medication Adherence Questionnaire | Six Months
  The SMAQ questionnaire was validated between 1998 and 1999 in Spanish population was treated with unboosted nelfinavir in patients with renal transplantation.
  It is a questionnaire to assess adherence to treatment consisting of 6 self-applied questions investigating different aspects of the phenomenon: a) oversights ; b ) times ; c ) adverse effects; d ) failure of the weekend ; e) quantification in the last week , and f ) quantification in the last quarter.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided